CLINICAL TRIAL: NCT03678246
Title: Low Skill Fibreoptic Glottis View in Obese Patients: Ramp vs Supine Sniffing Air Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2017-2135
Record Dates: First submitted 2018-08-20; First posted 2018-09-19 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Supine Position

STUDY DESIGN:
Intervention Model Description: Ramped vs Supine position
Masking Description: Images are reviewed by two senior anaesthetists who is not directly involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- LSFOI (Ramped) (Experimental): LSFOI (Ramped)
  Interventions: Procedure: Ramped position; Procedure: Supine position
- LSFOI (Supine) (Active Comparator): LSFOI (Supine)
  Interventions: Procedure: Ramped position; Procedure: Supine position

INTERVENTIONS:
Procedure: Ramped position — LSFOI glottis view
Procedure: Supine position — LSFOI glottis view

SUMMARY:
Aims: The investigators are employing a feasibility study to determine whether fibreoptic view of the glottis (vocal cords) during low skill fibreoptic intubation (FOI) via a laryngeal mask airway (LMA) in obese and severely obese patients is appropriate and feasible for future full-scale research. Obese, and severely and morbidly patients in Asia are classed as body mass index (BMI) of ≥ 30, ≥35 and ≥40 kg/m2, respectively.

DETAILED DESCRIPTION:
Aims: The investigators are employing a feasibility study to determine whether fibreoptic view of the glottis (vocal cords) during low skill fibreoptic intubation (FOI) via a laryngeal mask airway (LMA) in obese and severely obese patients is appropriate and feasible for future full-scale research. Obese, and severely and morbidly patients in Asia are classed as body mass index (BMI) of ≥ 30, ≥35 and ≥40 kg/m2, respectively.

Hypothesis: The glottis view during low skill FOI in obese and severely obese patients (BMI ≥30, and BMI ≥35 <40 kg/m2) is better in the ramp than in the standard supine 'sniffing air' position. Low skill FOI is a term for FOI via an LMA.

Methodology: As a feasibility study, the investigators will recruit 18 adult patients scheduled for elective surgery in obese and severely obese patients requiring tracheal intubation. A non-randomized cross over design in selected. The investigators will assess acceptability, implementation and practicality of such a study and also set criteria for success of this feasibility study.

Importance of proposed research: Obese patients present many anaesthetic challenges. The ramp position facilitates easier tracheal intubation and prolongs apnoea time. In cases of failed intubation, guidelines recommend insertion of an LMA to faciliate ventilation and oxygenation, allowing the option of low skill FOI to secure the airway. It may be performed in unanticipated difficult airway ('rescue' intubation after failed intubation by conventional techniques) and so may decrease patient morbidity and mortality. There is a knowledge gap regarding whether the glottis view during low skill FOI is superior in the ramp or standard supine sniffing position. It will help determine whether the study methodology and protocol needs modification and assess what changes may occur, before implementing a full-scale study. This will help form recommendations for future guidelines in difficult airway management.

Primary outcome is to measure feasibility of this study. The areas of focus addressed by this study are:

* the investigators will assess how many obese and severely obese patients we can recruit in the Pre-Operative Evaluation Clinic (PEC)

  1. Patient reaction and recruitment rate (accepting or declining invitation to the study)
  2. Patient dropout rate

     Integration: Previous studies evaluating FOI via the LMA have proved less straightforward than anticipated. Standard rostering of anaesthetic study members does not allocate the latter to the operating theatre where study patients are listed; this means the anaesthetic study team member needs to leave their own operating list elsewhere to deliver the study intervention leading to poor workflow. Also, the investigators used operating intubating fibrescopes, which had priority allocation to other (nonstudy) patients due to clinical reasons. In addition, the number of fibrescopes was greatly reduced due to maintenance and repair work. As such, our study protocol incorporates different workflows. As soon as a participant is recruited, the investigators will inform the roster consultant to allocate one of the anaesthetic study member to the operating theatre where a participant is listed to improve workflow. The investigators will also use grant funded disposable fibrescopes and grant funded fibrescope monitor.

     Assessment will be made of:
     1. Percentage of lists that contain study participants that have an allocated study team member, aiming for 80% allocation.
     2. Any workflow availability.

     Practicality: The investigators will assess for any difficulties when the patient is changed from a ramp to standard supine sniffing position by a coordinated team effort by theatre personnel.

     Secondary outcome measures will evaluate the technique of FOI via the LMA in our study population, comparing ramp and standard 'sniffing air' positions.
* Success of LMA insertion rate (after LMA insertion, an adequate capnography trace is obtained under study ventilation parameters, whilst in ramp position)
* LMA insertion times (time from picking up the LMA for insertion until adequate capnography trace is obtained, whilst in ramp position)
* Fibreoptic intubation times (time from picking up the fibrescope, after the patient has been place in the standard supine sniffing position, until adequate capnography trace is obtained)
* Airway manoeuvers to optimize glottis view
* Any complications

ELIGIBILITY:
Inclusion Criteria:

* obese and severely obese patients (BMI ≥30, and ≥35 but <40 kg/m2, respectively) undergoing elective bsurgery under general anaesthesia who require endotracheal intubation.

Exclusion Criteria:

* Morbidly obese patients (BMI ≥40 kg/m2)
* Patients with history of previous difficult endotracheal intubation
* Patients with two or more predictors of difficult face or laryngeal mask ventilation, or difficult intubation or the combination of both
* Mallamapatti score III-IV
* Interdental distance <3cm
* Thyromental distance <6cm
* Moderate to severe limitation of neck movement
* Previous head and neck radiotherapy or surgery
* Supraglottic lesion
* Patients with loose teeth
* Patients with ASA grade III (other than due to obesity) and grade IV are excluded from the study
* Patients needing a rapid sequence induction for rapid securement of the airway e.g. patients with symptoms of reflux (>1 episode per week), not starved as per standard nil by mouth guidelines, hiatus hernia, previous gastric surgery
* Pregnant women
* Patients below the age of 21 years old
* Patients unfit to give consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Feasibility study | 6 months
  patient recruitment rate and ability to complete the study

SECONDARY OUTCOMES:
Positioning challenges | 6 months
  descriptive scale with free text comments on difficulties encountered during positioning from ramped to supine
Success of LMA insertion rate | 6 months
  Success of LMA insertion rate with number of attempts stated
LMA insertion times | 6 months
  LMA insertion times
Fibreoptic intubation times | 6 months
  Fibreoptic intubation times
Airway manoeuvres to optimize glottis view | 6 months
  options include jaw thrust and withdrawal of LMA
Any complications | 6 months
  descriptive scale listing the problems/complications encountered during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore